CLINICAL TRIAL: NCT02607605
Title: A Prospective, Observational Trial on the Diagnostic and Prognostic Value of Cell-free DNA in Advanced Lung Cancer With Leptomeningeal Metastases
Brief Title: A Prospective, Observational Trial on the Diagnostic and Prognostic of LM
Acronym: ctDNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li-kun Chen, associate professor, Sun Yat-sen University
Other Study IDs: 201507004
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Lung Neoplasms; Meningeal Carcinomatosis
Keywords: lung cancer; leptomeningeal metastases; cell-free DNA
MeSH Terms: conditions — Lung Neoplasms; Meningeal Carcinomatosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — patient's cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary purpose of this study is to compare the positive rate between the cell-free DNA and cytological examination of cerebrospinal fluid in Advanced lung cancer with leptomeningeal metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who was confirmed primary lung cancer by pathologic histology or cytology
2. Adult patients (≥18 years and ≤75 years). ECOG Performance Status 0 or 1.Life expectancy of at least 12 weeks.
3. Clinical symptoms and imaging tests are highly suspicious of advanced lung cancer with leptomeningeal metastases
4. Without contraindications to lumbar puncture

Exclusion Criteria:

1. Patients who have primary benign or malignant brain tumor and metastatic malignant brain tumor
2. Patients who have contraindications to lumbar puncture
3. Serious uncontrolled systemic disease including active infection,uncontrolled hypertension,diabetes,unstable angina,congestive heart failure,myocardial infarction,severe arrhythmia which needs drugs,hepatic、renal and metabolic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical symptoms and imaging tests are highly suspicious of advanced lung cancer with leptomeningeal metastases
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2015-08; Primary Completion 2019-12 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
positive rate between the cell-free DNA and cytological examination of cerebrospinal fluid | 2 years

SECONDARY OUTCOMES:
The relationship between the number of cell-free DNA and OS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: li-kun Chen, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University of cancer center, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Pan W, Gu W, Nagpal S, Gephart MH, Quake SR. Brain tumor mutations detected in cerebral spinal fluid. Clin Chem. 2015 Mar;61(3):514-22. doi: 10.1373/clinchem.2014.235457. Epub 2015 Jan 20. PMID 25605683
- [Result] Newman AM, Bratman SV, To J, Wynne JF, Eclov NC, Modlin LA, Liu CL, Neal JW, Wakelee HA, Merritt RE, Shrager JB, Loo BW Jr, Alizadeh AA, Diehn M. An ultrasensitive method for quantitating circulating tumor DNA with broad patient coverage. Nat Med. 2014 May;20(5):548-54. doi: 10.1038/nm.3519. Epub 2014 Apr 6. PMID 24705333